CLINICAL TRIAL: NCT04095065
Title: The Intersection of Alcohol and Sex: Engineering an Online STI Prevention Program
Brief Title: Engineering an Online STI Prevention Program: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: University of North Carolina, Greensboro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: R01AA02931-3
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Consumption; Sexually Transmitted Diseases
Keywords: Multiphase optimization strategy (MOST); College students
MeSH Terms: conditions — Alcohol Drinking; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- itMatters (Experimental): Participants will have access to content focused on general knowledge and injunctive and descriptive norms for a period up to 3 weeks.
  Interventions: Behavioral: itMatters
- itMatters and itMatters Sexual Violence Prevention (Experimental): Participants will have access to content focused on general knowledge and injunctive and descriptive norms related to alcohol use and sex. Additionally, participants will have access to content focused on sexual violence including basic information and bystander intervention. This content will be available for a period up to 3 weeks.
  Interventions: Behavioral: itMatters and itMatters Sexual Violence Prevention
- itMatters Well-being and itMatters Sexual Violence Prevention (Experimental): Participants will have access to content focused on basic information related to sleep wellness and time management. In Addition, participants will have access to content focused on sexual violence including basic information and bystander intervention. This content will be available for a period up to 3 weeks.
  Interventions: Behavioral: itMatters Well-being and itMatters Sexual Violence Prevention
- itMatters Well-being (Experimental): Participants will have access to content focused on basic information related to sleep wellness and time management. This content will be available for a period up to 3 weeks.
  Interventions: Behavioral: itMatters Well-being

INTERVENTIONS:
Behavioral: itMatters — Increase knowledge related to STIs, STI risk, alcohol impairment, condom use, alcohol use behavior tracking skill, testing & treatment knowledge. Correct misperceptions regarding approval (injunctive norms) and prevalence (descriptive norms) of alcohol misuse & sexual risk taking.
  Arms: itMatters
Behavioral: itMatters and itMatters Sexual Violence Prevention — Increase knowledge related to STIs, STI risk, alcohol impairment, condom use, alcohol use behavior tracking skill, testing & treatment knowledge. Correct misperceptions regarding approval (injunctive norms) and prevalence (descriptive norms) of alcohol misuse & sexual risk taking. Additionally, increased knowledge related to sexual violence (prevalence, key definitions, individual rights and responsibilities, laws) and increased knowledge, efficacy, and intentions to use bystander behaviors during moments of sexual violence.
  Arms: itMatters and itMatters Sexual Violence Prevention
Behavioral: itMatters Well-being and itMatters Sexual Violence Prevention — Increase knowledge related to sleep, including biological effects of sleep and sleep hygiene. Increase knowledge related to time management, including important definitions, sleep management strategies, and effective time management routines. Additionally, increased knowledge related to sexual violence (prevalence, key definitions, individual rights and responsibilities, laws) and increase knowledge, efficacy, and intentions to use bystander behaviors during moments of sexual violence.
  Arms: itMatters Well-being and itMatters Sexual Violence Prevention
Behavioral: itMatters Well-being — Increase knowledge related to sleep, including biological effects of sleep and sleep hygiene. Increase knowledge related to time management, including important definitions, sleep management strategies, and effective time management routines.
  Arms: itMatters Well-being

SUMMARY:
The overall objective of the proposed research is to reduce the incidence of sexually transmitted infections (STIs) among college students. The investigators propose to accomplish this by using the innovative, engineering-inspired multiphase optimization strategy (MOST) to develop a highly effective, appealing, economical, and readily scalable internet-delivered behavioral intervention targeting the intersection of alcohol use and sexual risk behavior. The rate of STIs on college campuses is alarming: one in four college students is diagnosed with an STI at least once during their college experience. Sexual activity when drinking alcohol is highly prevalent among college students. Alcohol use is known to contribute to the sexual risk behaviors that are most responsible for the transmission of STIs, namely unprotected sex, contact with numerous partners, and "hook-ups" (casual sexual encounters). Few interventions have been developed that explicitly target the intersection of alcohol use and sexual risk behaviors, and none have been optimized. In order to reduce the incidence of STI transmission among this and other high-risk groups, a new approach is needed. MOST is a comprehensive methodological framework that brings the power of engineering principles to bear on optimization of behavioral interventions. MOST enables researchers to experimentally test the individual components in an intervention to determine their effectiveness, indicating which components need to be revised and re-tested. Given the high rates of alcohol use and sex among college students, the college setting provides an ideal opportunity for intervening on alcohol use and sexual risk behaviors. The proposed study will include a diverse population of college students on 4 campuses which will increase the generalizability of the findings. The specific aims are to (1) develop and pilot test an initial set of online intervention components targeting the link between alcohol use and sexual risk behaviors, (2) use the MOST approach to build an optimized preventive intervention, and (3) evaluate the effectiveness of the newly optimized preventive intervention using a fully powered randomized controlled trial (RCT). This work will result in a new, more potent behavioral intervention that will reduce the incidence of STIs among college students in the US, and will lay the groundwork for a new generation of highly effective STI prevention interventions aimed at other subpopulations at risk.

DETAILED DESCRIPTION:
As part of the MOST approach, the investigators have conducted two optimization trials (NCT02897804 and NCT 03408743) to identify the optimized intervention. The current study is the randomized controlled trial of the optimized intervention.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled at an American college or University
* A first-year college student
* 18 years or older
* Have not gone through previous versions of itMatters

Exclusion Criteria:

* Not a first year student or transfer student
* Younger than 18 years old
* Have gone through previous versions of itMatters

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3098 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Unprotected behavior at most recent vaginal or anal sex collected via online questionnaire | Condom use will be assessed 60 days post-intervention.
  Two items ask whether or not a condom was used for vaginal or anal sex, for those who indicated recently having vaginal or anal sex. The variables will be reported as prevalence of this behavior and likely used as a dichotomous variable (unprotected/protected) in regression analyses.
Penetrative sex at most recent hookup collected via online questionnaire | This measure will be assessed 60 days post-intervention
  This item asks whether or not the most recent hookup included vaginal or anal sex. This will be reported as prevalence of the behavior and likely used as a dichotomous variable in regression analyses.
Attitudes about sexual violence | This measure will be assessed 60 days post-intervention.
  Four items ask about perceptions of sexual violence, including language, consent, pressure, and inappropriate touching. The scale will reflect the average perceptions of sexual violence attitudes.

SECONDARY OUTCOMES:
Injunctive norms about the intersection of alcohol and sex | This measure will be assessed 60 days post-intervention.
  This scale consists of 5 items reflecting the average perceived approval of the alcohol and sex behaviors, ranging from strongly disapprove to strongly approve.
Descriptive norms about the intersection of alcohol and sex | This measure will be assessed 60 days post-intervention.
  This scale consists of 5 items reflecting the average perceived prevalence of the alcohol and sex behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Linda M Collins, PhD, Principal Investigator — Penn State University
Locations (4):
- United States (4):
  - Fresno State University, Fresno, California
  - University of North Carolina - Greensboro, Greensboro, North Carolina
  - North Dakota State University, Fargo, North Dakota
  - Middle Tennessee State University, Murfreesboro, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanner AE, Guastaferro KM, Rulison KL, Wyrick DL, Milroy JJ, Bhandari S, Thorpe S, Ware S, Miller AM, Collins LM. A Hybrid Evaluation-Optimization Trial to Evaluate an Intervention Targeting the Intersection of Alcohol and Sex in College Students and Simultaneously Test an Additional Component Aimed at Preventing Sexual Violence. Ann Behav Med. 2021 Nov 18;55(12):1184-1187. doi: 10.1093/abm/kaab003. PMID 33704366